CLINICAL TRIAL: NCT05260749
Title: Real-time fMRI Neurofeedback Training on the Anterior Insula Via Interoceptive Processing and Its Behavioral Effects
Brief Title: Real-time fMRI Neurofeedback Training on the Anterior Insula Based on Interoceptive Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Shuxia Yao, Associate Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-85
Record Dates: First submitted 2022-02-08; First posted 2022-03-02 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: real-time neurofeedback; anterior insula; Interoceptive Processing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neurofeedback training (Experimental): Subjects in the neurofeedback training group are instructed to regulate their anterior insula activity based on the visual neurofeedback.
  Interventions: Procedure: real-time fMRI neurofeedback training procedure
- Sham control1 (Sham Comparator): Subjects in the sham control group receive the same instruction but perform the regulation based on neurofeedback from a whole slice of top brain (a controlled sham region).
  Interventions: Procedure: real-time fMRI sham-controlled neurofeedback training procedure
- Sham control2 (Sham Comparator): Subjects in the sham control group receive the same instruction but perform the regulation based on neurofeedback from the middle temporal gyrus (a controlled sham region).
  Interventions: Procedure: real-time fMRI sham-controlled neurofeedback training procedure

INTERVENTIONS:
Procedure: real-time fMRI neurofeedback training procedure — real-time fMRI neurofeedback training procedure running on the Turbo Brain voyager (TBV) 3.2 software (Brain Innovation, Maastricht, The Netherlands)
  Arms: Neurofeedback training
Procedure: real-time fMRI sham-controlled neurofeedback training procedure — real-time fMRI sham neurofeedback training procedure running on the Turbo Brain voyager (TBV) 3.2 software (Brain Innovation, Maastricht, The Netherlands)
  Arms: Sham control1; Sham control2

SUMMARY:
The main aim of the study is to investigate whether subjects can learn self control of activity of the anterior insula via real-time functional magnetic resonance imaging (fMRI) neurofeedback training based on a regulation strategy of interoceptive processing.

DETAILED DESCRIPTION:
A double-blinded, placebo-controled, between-subject design is employed in this study. In a randomized order, a total of 90 healthy subjects will be recruited and assigned into the experimental group (EG; N=33), which receives real feedback from the left anterior insula, or the control group (CG; N=33) which receives sham feedback from a whole slice of top brain, or the control group 2 (CG2; N=33) wich receives sham feedback from the middle temporal gyrus. Neurofeedback training consists of 4 training sessions with real-time feedback and 1 transfer session without feedback. A heartbeat detection task pre- and post-training was used to determine interoceptive accuracy changes induced by neurofeedback training. A pre-training empathy task before training was used to localise the anterior insula and as a baseline of empathic response. A post-training empathy task was used to determine the effects of neurofeedback training on empathic response by comparing with the pre-training one. Behavioral and fMRI data are collected during the empathy tasks and the neurofeedback task. Personality traits of subjects are assessed using validated Chinese version questionnaires, including the Toronto Alexithymia Scale (TAS), Multidimensional Assessment of Interoceptive Awareness (MAIA), Interoceptive Confusion Questionnaire (ICQ), Beck Depression Inventory (BDI), State-Trait Anxiety Inventory (STAI), Autism Spectrum Quotient (ASQ), Empathy Quotient (EQ). Subjects are asked to complete Positive and Negative Affect Schedule (PANAS) twice before and after the neurofeedback training task.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any past or present psychiatric or neurological disorders

Exclusion Criteria:

* History of brain injury Medical or mental illness

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Neural activity of the anterior insula based on blood oxygen level-dependent (BOLD) signal | 1 hour
  The anterior insula activity induced by neurofeedback training relative to sham feedback training

SECONDARY OUTCOMES:
Confidence rating scores of interoceptive sensitivity | 1 hour
  Subjects are asked to rate to what extent they can feel their heartbeat based on a Likert Scale ranging from 1-9 (1 = very low and 9 = very high)
pain empathy ratings scores | 1 hour
  Subjects were required to rate their empathic feeling towards painful pictures on a Likert Scale ranging from 1-9 (1 = not at all and 9 = very painful) before and after neurofeedback training.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Shuxia, Dr, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China(UESTC), Chengdu, Sichuan, China

REFERENCES:
- [Derived] Zhang Y, Zhang Q, Wang J, Zhou M, Qing Y, Zou H, Li J, Yang C, Becker B, Kendrick KM, Yao S. "Listen to your heart": A novel interoceptive strategy for real-time fMRI neurofeedback training of anterior insula activity. Neuroimage. 2023 Dec 15;284:120455. doi: 10.1016/j.neuroimage.2023.120455. Epub 2023 Nov 10. PMID 37952779